CLINICAL TRIAL: NCT06372548
Title: The Effect of Cognitive Appraisal Theory on Adherence in Rehabilitation Training Games for Children With Amblyopia
Brief Title: Rehabilitation Training Games for Children With Amblyopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhu Dian (Other)
Responsible Party: Sponsor-Investigator, Zhu Dian, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NEADS0004
Record Dates: First submitted 2024-03-24; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Amblyopia; Amblyopia Occlusion; Child Behavior; Adherence, Treatment
MeSH Terms: conditions — Amblyopia; Child Behavior; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Find You! Cure My Animal Friends (Experimental): Participants in the experimental group completed the game in this app. The goal of the game is to guide the amblyopic children to develop the habit of rehabilitation training, so that the amblyopic children will keep their interest in completing the exercises according to the time in the game. A story of an animal intern doctor is constructed, and the player will play the role of an animal doctor according to the guidance of the plot, wear the corresponding eye patches and complete the set visual training tasks in the game. The study aims to improve the overall treatment adherence by increasing the attractiveness of the visual training game to children, cultivating long-term training habits, and mitigating the negative effects of amblyopia treatment. The path to achieve this goal consists of the following components: (1) narrative content, (2) interactive forms combined with masking therapy, (3) incentives, and (4) visual design that is consistent with children's preferences.
  Interventions: Device: Find You! Cure My Animal Friends
- DuoBao Vision Training System (Active Comparator): Software Co.'s DuoBao Vision Training System. A number of visual function tests and ophthalmology strabismus amblyopia specialist examinatio. The data is transmitted to the data center and the expert intelligent system to develop a targeted personalized amblyopia training program. Control group participants completed the training components in this app.
  Interventions: Device: DuoBao Vision Training System

INTERVENTIONS:
Device: Find You! Cure My Animal Friends — Introduced cognitive evaluation theory combined with masking therapy to develop a gamified product that guides amblyopic children to develop habits for the purpose of rehabilitation training.
  Arms: Find You! Cure My Animal Friends
Device: DuoBao Vision Training System — This is a visual training app where participants are required to complete several training tasks.
  Arms: DuoBao Vision Training System

SUMMARY:
A gamification product was developed to guide children with amblyopia to develop rehabilitation training habits by combining cognitive evaluation theory and occlusion therapy. A randomized controlled trial was conducted to examine the ease of use, acceptability and treatment compliance of the game.

DETAILED DESCRIPTION:
The experimental group was subjected to a 20-minute daily, 4-week intervention experiment, which included a story background on the start page, eye patches to be put on according to the guidelines, fine eye training, and visual stimulation training, with short breaks between the different modes. The control group was given an experimental intervention using a competing product, with the same duration and format as the experimental group. After completion of the intervention, the participating children completed the MMAS-8 adherence scale with the help of their parents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of amblyopia (including refractive amblyopia, strabismic amblyopia and mixed).
* The child has no significant IQ deficits and has no difficulty communicating with others.
* The children's teachers and parents gave their informed consent to participate in the experiment. The informed consent form was signed by the parents and is shown in the Appendix.

Exclusion Criteria:

* Severe amblyopia.
* Suffering from other psychological or physical disorders.
* Parents did not agree to sign the informed consent form or the child was not willing to participate in this experiment.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
8-Item Morisky Medication Adherence Scale (MMAS-8): | baseline and study completion (after 8 weeks)
  A patient's adherence to therapy can be evaluated using the eight-question Morisky Medication Adherence Scale-8 (MMAS-8).The total score of the MMAS-8 scale is the sum of the scores of the above 8 questions, and the score range is 0~8. Higher scores indicate better medication adherence. 8 indicates good adherence; 6~7 indicates moderate adherence; <6 indicates poor adherence.

SECONDARY OUTCOMES:
User Experience Questionnaire (UEQ) | study completion (after 8 weeks)
  Enabling prompt and accurate user experience measurement is the primary goal of the UEQ.UEQ was administered post-experiment to swiftly and accurately measure user experience. Covering 26 items across six domains, UEQ evaluated the impact of the amblyopia rehabilitation training product on both children and their parents. Due to its language complexity, the questionnaire was completed with parental assistance.1 for disagree, 7 for strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Dian Zhu, Dr, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No